CLINICAL TRIAL: NCT05286528
Title: Retrospective, Non-interventional Study to Evaluate Chronic Myeloid Leukemia Treatment Landscape and Real-life Treatment Outcomes in Hungary: Analysis of National Health Insurance Fund Database
Brief Title: Study to Evaluate Chronic Myeloid Leukemia Treatment Landscape and Real-life Treatment Outcomes in Hungary: Analysis of National Health Insurance Fund Database
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1871064
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Results first posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Chronic Myeloid Leukaemia
Keywords: tyrosine kinase inhibitor (TKI)
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — bosutinib; Imatinib Mesylate; nilotinib; Dasatinib; ponatinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Bosutinib — Bosutinib as prescribed in real world
Drug: Imatinib — Imatinib as prescribed in real world
Drug: Nilotinib — Nilotinib as prescribed in real world
Drug: Dasatinib — Dasatinib as prescribed in real world
Drug: Ponatinib — Ponatinib as prescribed in real world

SUMMARY:
The objectives of this study are to describe patient demographics, clinical and disease characteristics and treatment patterns of Chronic Lymphoid Leukaemia (CML) in Hungary.

The primary endpoint of this study is the overall survival of CML patients treated with tyrosine kinase inhibitors in Hungary. The Overall Survival (OS) of all enrolled patients, OS by sequence pattern and by the number of treatment lines will be analyzed.

Secondary objectives are description of the treatment length in 1st and later lines, incidence and prevalence of CML, the patient demographics (as age, gender, comorbidities), average number of patients' comorbidities, most frequent comorbidities and patient number with comorbidities at baseline and at different treatment lines by investigated Thyrosine Kinase Inhibitor (TKI), distribution of the investigated TKI therapies by treatment lines

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients diagnosed with chronic myeloid leukemia
* Patients receiving tyrosine kinase inhibitor therapy under the terms of the current marketing authorization

Exclusion Criteria:

* Patients receiving TKI for non-CML diagnoses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All CML patients treated with any TKI with CML diagnosis based on the International Classification of Diseases - 10th revision (ICD) during the investigated timeframe
Sampling Method: Non-Probability Sample
Enrollment: 1484 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants, who received tyrosine kinase inhibitors (imatinib, dasatinib, nilotinib, bosutinib, or ponatinib) anytime from 01 January 2009 to 30 June 2020, under the terms of the current marketing authorization, inclusion criteria, for treatment of chronic myeloid leukemia (CML), was retrieved from database National Health Insurance Fund (NHIF) of Hungary.
Groups:
- Participants With CML: Participants who received their first tyrosine kinase inhibitors (imatinib, dasatinib, nilotinib, bosutinib or ponatinib) to treat CML (from 01 January 2011 - 30 June 2020) under standard real world clinical practice in Hungary (under the terms of the current marketing authorization). Data collection started 2 years before (01 January 2009), as reference years in order to detect only the real starting therapies from 2011.
Period: Overall Study
Arm/Group | Participants With CML
Started | 1484
Completed | 1484
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis set included all participants treated with tyrosine kinase inhibitors based on chronic myeloid leukemia diagnosis between 01 January 2009 to 30 June 2020.
Arm/Group | Participants With CML
Number analyzed (Participants) | 1484
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.14 (17.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 704
  Male | 780
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Rate: All Participants
Description: Overall survival rate in this study was defined as percentage of participants alive during analysis period of 01-January-2011 till 30-June-2020. 5 years overall survival rate was demonstrated with Kaplan-Meier curve.
Time Frame: 5 years, during analysis period from 01-January-2011 till 30-June-2020 (retrieved data assessed in this observational study for approximately 1.2 years)
Population: Analysis set included all participants initiated with first line tyrosine kinase inhibitors based on chronic myeloid leukemia diagnosis between 01 January 2011 to 30 June 2020.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With CML
Number analyzed (Participants) | 1484
Percentage of participants | 77.1

2. Primary Outcome: Overall Survival Rate: Type of First Line TKI
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With CML
Number analyzed (Participants) | 1484
Percentage of participants | 77.1

3. Primary Outcome: Overall Survival Rate: Type of Second Line TKI
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Analysis set included all participants initiated with second line tyrosine kinase inhibitors based on chronic myeloid leukemia diagnosis between 01 January 2011 to 30 June 2020. Here, Overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Groups:
- Participants With CML: Participants who received their second tyrosine kinase inhibitors (imatinib, dasatinib, nilotinib, bosutinib or ponatinib) to treat CML (from 01 January 2011 - 30 June 2020) under standard real world clinical practice in Hungary (under the terms of the current marketing authorization). Data collection started 2 years before (01 January 2009), as reference years in order to detect only the real starting therapies from 2011.
Arm/Group | Participants With CML
Number analyzed (Participants) | 647
Percentage of participants | 71.5

4. Primary Outcome: Overall Survival Rate: Per Sequence of Treatment
Description: as for outcome 1
Time Frame: as for outcome 1
Population: NHIF did not provide data for event below 10 participants. Apart from 2 sequences all rest sequences had low yearly participants during the whole studied period (less than 10 participants). Hence data for analysis for Overall Survival rate by sequence was not collected and analyzed for whole population.
Arm/Group | Participants With CML
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not collected for the study
Description: Due to non-interventional nature of study, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not meet, hence adverse events were not collected and reported.
Arm/Group | Participants With CML
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT05286528/Prot_SAP_000.pdf